CLINICAL TRIAL: NCT06746935
Title: Reconstruction of Deficient Atrophic Ridges Using Guided Bone Regeneration Technique With Native Collagen Membrane and Polytetrafluoroethylene Membrane (Randomized Clinical Trial)
Brief Title: Reconstruction of Deficient Atrophic Ridges Using Guide Bone Regeneration Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohannad Ahmed Ismail, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0001-6142-0568
Record Dates: First submitted 2024-12-15; First posted 2024-12-24 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Ridge Augmentation; Bone Augmentation
Keywords: ridge augmentation; Polytetrafluoroethylene; native collagen membrane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patients were randomly allocated into two groups utilizing Random Allocation Software version 2.0. then the allocation was concealed in opaque sealed envelopes. In both groups. The allocation was revealed to the operator just before the surgery. On the other hand, the patients, outcome assessor and the statistician who analyzed the collected data and performed the statistical analysis were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group B polytetrafluoroethylene membrane. (Active Comparator): Particulate bone mixture 1:1 autogenous and xenogenic bone covered with polytetrafluoroethylene membrane.
  Interventions: Procedure: Polytetrafluoroethylene membrane.
- Study Group A native collagen membrane. (Experimental): Particulate bone mixture 1:1 autogenous and xenogenic bone covered with native collagen membrane.
  Interventions: Procedure: Collagen membrane.

INTERVENTIONS:
Procedure: Collagen membrane. — Particulate bone mixture 1:1 autogenous and xenogenic bone covered with native collagen membrane.
  Arms: Study Group A native collagen membrane.
Procedure: Polytetrafluoroethylene membrane. — Particulate bone mixture 1:1 autogenous and xenogenic bone covered with polytetrafluoroethylene membrane.
  Arms: Control Group B polytetrafluoroethylene membrane.

SUMMARY:
patients will be informed of the nature of the research work and informed consent will be obtained then randomized in 2 groups. Mixture 1:1 autogenous and xenogenic bone covered with Polytetrafluoroethylene membrane control group and study group p covered with native collagen membrane.

* Patients of both groups will be subjected to CBCT (diagnostic for upper arch), diagnostic wax-up and stent fabrication.
* Intra operative procedures (for both groups) followed by CBCT will be taken for every patient after 4 months.

Both the study and control group will receive:

* In Recipient site, using 15C blade on Bard Parker handle incision of full thickness mucoperiosteal flap inorder to obtain, three-line pyramidal flap, reflection using mucoperiosteal elevator molt 9.
* The defective site is reevaluated after its primary evaluation on CBCT using UNC (University of North Carolina) periodontal probe and a template is cut using sterile suture pack, prior to donor site preparation.
* Flap advancement using periosteal releasing incision inorder to allow later tension free flap closure.
* In Donor site, mucoperiosteal flap is done, auto chip maker (ACM) is used for autogenous bone harvesting.
* Autogenous particulate bone graft is obtained using auto chip maker bur (ACM), in implant contra 20:1 using surgical motor recommended drilling speed 100 rpm and maximum torque 50 Ncm. as well as, using bone scrapper in push direction.
* Xenogenic bone graft particles (De-proteinized bovine bone mineral small granules (0.25-1 mm). is added to the autogenous bone particles to obtain homogenous mixture ratio 1:1.
* The gold standard is a mixture of autogenous bone containing viable cells and xenogenic bone which has slower rate of resorption is to be placed in recipient decorticated site and covered by PTFE membrane.
* The assemble is to be fixed by titanium bone tacks of diameter 2.5 mm and length 3.5 mm, to avoid micro movements of particulate bone assembly.
* In the Study group: The assemble is going to be covered by resorbable collagen membrane and fixed by tacks.
* Recheck adequate flap advancement by visualizing passive flap approximation, to allow tension free closure.
* Double line closure using horizontal mattress placed 5mm away from flap margins followed by interrupted sutures on top to allow contact area which is preferred to point contact and wound edge eversion.

DETAILED DESCRIPTION:
.General operative procedures The selected patients will be informed of the nature of the research work and informed consent will be obtained then randomized in equal proportions between control group particulate bone mixture 1:1 autogenous and xenogenic bone covered with Polytetrafluoroethylene membrane and study group particulate bone mixture 1:1 autogenous and xenogenic bone covered with native collagen membrane.

* Patients of both groups will be subjected to CBCT (diagnostic for upper arch), diagnostic wax-up and stent fabrication.
* Intra operative procedures (for both groups) followed by CBCT will be taken for every patient after 4 months.
* Infiltration local anesthesia will be given to the patient (Articaine 4% 1:100 000 epinephrine).

Both the study and control group will receive:

* In Recipient site, preparation 1st to obtain, three-line pyramidal flap.
* Flap advancement using periosteal releasing incision.
* In Donor site, auto chip maker (ACM) is used for autogenous bone harvesting and xenogenic bone graft particles mixture ratio 1:1.
* The assemble is to be fixed by titanium bone tacks. In the Study group: The assemble is going to be covered by collagen membrane.
* Double line closure using horizontal mattress placed 5mm away from flap margins followed by interrupted sutures on top to allow contact area which is preferred to point contact and wound edge eversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with maxillary residual alveolar bone height not less than 8 mm.
* Alveolar bone width from less than or equal 5 mm.
* Both sexes.
* At least missing single tooth.
* Previous Failed Implants.
* Previous Failed Grafting.

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with bone disease that may affect normal healing, example; hyperparathyroidism.
* Patients had radiotherapy and chemotherapy in head and neck.
* Patients had neoplasms in sites to be grafted.
* Patients with Metabolic diseases uncontrolled diabetic patients, Glycated hemoglobin (Hb A1c) more than 7 mg\dl.

Ages: 20 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
Quantity of bone gain. | After 4 months from ridge augmentation.
  Measured using linear measurements from Cone Beam Computed Tomography (CBCT) in millimeters (mm).

SECONDARY OUTCOMES:
Soft tissue dehiscence. | Starting from Week 1. Binary Yes or No.
  Exposure of barrier membrane and impaied wound healing.

OTHER OUTCOMES:
Pain assessment. | Day 1.
  Location,onset and character. Using questionnaire. Using Visual Analogue Scale. Numerical from 0 to 10. 0 no pain and 10 the worst pain.
  * Numerical from 0 to 10. Questionnaire.
  * Numerical from 0 to 10.
  * Questionnaire.
  * Numerical from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. Youssef, PHD., Study Director — Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Cairo University, Egypt
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammerle CH, Jung RE. Bone augmentation by means of barrier membranes. Periodontol 2000. 2003;33:36-53. doi: 10.1046/j.0906-6713.2003.03304.x. No abstract available. PMID 12950840
- [Background] Pellegrino G, Lizio G, Corinaldesi G, Marchetti C. Titanium Mesh Technique in Rehabilitation of Totally Edentulous Atrophic Maxillae: A Retrospective Case Series. J Periodontol. 2016 May;87(5):519-28. doi: 10.1902/jop.2016.150432. Epub 2016 Jan 12. PMID 26759078
- [Background] Polis-Yanes C, Cadenas-Sebastian C, Gual-Vaques P, Ayuso-Montero R, Mari-Roig A, Lopez-Lopez J. Guided Bone Regeneration of an Atrophic Maxilla Using Heterologous Cortical Lamina. Case Rep Dent. 2019 Jun 11;2019:5216362. doi: 10.1155/2019/5216362. eCollection 2019. PMID 31308978
- [Background] Jensen J, Sindet-Pedersen S. Autogenous mandibular bone grafts and osseointegrated implants for reconstruction of the severely atrophied maxilla: a preliminary report. J Oral Maxillofac Surg. 1991 Dec;49(12):1277-87. doi: 10.1016/0278-2391(91)90303-4. PMID 1955919
- [Background] Misch CM. Comparison of intraoral donor sites for onlay grafting prior to implant placement. Int J Oral Maxillofac Implants. 1997 Nov-Dec;12(6):767-76. PMID 9425757
- [Background] Montazem A, Valauri DV, St-Hilaire H, Buchbinder D. The mandibular symphysis as a donor site in maxillofacial bone grafting: a quantitative anatomic study. J Oral Maxillofac Surg. 2000 Dec;58(12):1368-71. doi: 10.1053/joms.2000.18268. PMID 11117684
- [Background] Gungormus M, Yavuz MS. The ascending ramus of the mandible as a donor site in maxillofacial bone grafting. J Oral Maxillofac Surg. 2002 Nov;60(11):1316-8. doi: 10.1053/joms.2002.35731. PMID 12420267
- [Background] Clavero J, Lundgren S. Ramus or chin grafts for maxillary sinus inlay and local onlay augmentation: comparison of donor site morbidity and complications. Clin Implant Dent Relat Res. 2003;5(3):154-60. doi: 10.1111/j.1708-8208.2003.tb00197.x. PMID 14575631
- [Background] Pourabbas R, Nezafati S. Clinical results of localized alveolar ridge augmentation with bone grafts harvested from symphysis in comparison with ramus. J Dent Res Dent Clin Dent Prospects. 2007 Spring;1(1):7-12. doi: 10.5681/joddd.2007.002. Epub 2007 Jun 10. PMID 23277827
- [Background] Acocella A, Bertolai R, Colafranceschi M, Sacco R. Clinical, histological and histomorphometric evaluation of the healing of mandibular ramus bone block grafts for alveolar ridge augmentation before implant placement. J Craniomaxillofac Surg. 2010 Apr;38(3):222-30. doi: 10.1016/j.jcms.2009.07.004. Epub 2009 Aug 3. PMID 19648020
- [Background] Spin-Neto R, Landazuri Del Barrio RA, Pereira LA, Marcantonio RA, Marcantonio E, Marcantonio E Jr. Clinical similarities and histological diversity comparing fresh frozen onlay bone blocks allografts and autografts in human maxillary reconstruction. Clin Implant Dent Relat Res. 2013 Aug;15(4):490-7. doi: 10.1111/j.1708-8208.2011.00382.x. Epub 2011 Aug 11. PMID 21834864
- [Background] Acocella A, Bertolai R, Ellis E 3rd, Nissan J, Sacco R. Maxillary alveolar ridge reconstruction with monocortical fresh-frozen bone blocks: a clinical, histological and histomorphometric study. J Craniomaxillofac Surg. 2012 Sep;40(6):525-33. doi: 10.1016/j.jcms.2011.09.004. Epub 2011 Nov 9. PMID 22075326
- [Background] Dasmah A, Thor A, Ekestubbe A, Sennerby L, Rasmusson L. Particulate vs. block bone grafts: three-dimensional changes in graft volume after reconstruction of the atrophic maxilla, a 2-year radiographic follow-up. J Craniomaxillofac Surg. 2012 Dec;40(8):654-9. doi: 10.1016/j.jcms.2011.10.032. Epub 2011 Dec 3. PMID 22137760
- [Background] AlGhamdi AS. Post-surgical complications of symphyseal block graft with and without soft tissue grafting. Saudi Med J. 2013 Jun;34(6):609-15. PMID 23756926
- [Background] Hernandez-Alfaro F, Sancho-Puchades M, Guijarro-Martinez R. Total reconstruction of the atrophic maxilla with intraoral bone grafts and biomaterials: a prospective clinical study with cone beam computed tomography validation. Int J Oral Maxillofac Implants. 2013 Jan-Feb;28(1):241-51. doi: 10.11607/jomi.2405. PMID 23377071
- [Background] Monje A, Monje F, Chan HL, Suarez F, Villanueva-Alcojol L, Garcia-Nogales A, Wang HL. Comparison of microstructures between block grafts from the mandibular ramus and calvarium for horizontal bone augmentation of the maxilla: a case series study. Int J Periodontics Restorative Dent. 2013 Nov-Dec;33(6):e153-61. doi: 10.11607/prd.1664. PMID 24116370
- [Background] Aloy-Prosper A, Penarrocha-Oltra D, Penarrocha-Diago M, Penarrocha-Diago M. The outcome of intraoral onlay block bone grafts on alveolar ridge augmentations: a systematic review. Med Oral Patol Oral Cir Bucal. 2015 Mar 1;20(2):e251-8. doi: 10.4317/medoral.20194. PMID 25662543
- [Background] Reininger D, Cobo-Vazquez C, Monteserin-Matesanz M, Lopez-Quiles J. Complications in the use of the mandibular body, ramus and symphysis as donor sites in bone graft surgery. A systematic review. Med Oral Patol Oral Cir Bucal. 2016 Mar 1;21(2):e241-9. doi: 10.4317/medoral.20938. PMID 26827063
- [Background] Khoury F: Augmentation of severe bony defects with intraoral bone grafts: biological approach and long-term results J Oral Maxillo Fac Surg 2017Volume 46, Supplement 1, Pages 26-27.
- [Background] Claudino M, Julio C L, Luis E M, Bernardo M, Fernando G, tomographic evaluation of atrophic maxilla rehabilitated with autogenous and xenogeneic block grafts. Journal of Research in Dentistry 2017, 4(4):112-117.